CLINICAL TRIAL: NCT01388907
Title: Efficacy and Safety of Prevadh™ in the Prevention of Adhesions in Gynaecological Surgery: a Multicenter, Randomized, French Study
Brief Title: Efficacity Assessment of PREVADH® in Adhesion Prevention in Gynaecologic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Collaborators: Registrat-Mapi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLI 9821-2
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Results first posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Uterine Fibroids; Fertility Disorders
Keywords: myomectomy; adhesion prevention; pregnancy rate
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevadh film (Experimental): Patient randomized in this arm have been treated with Prevadh film applied on the uterine surgical sites, at the end of the myomectomy surgery to prevent post-surgey adhesion formation.
  Interventions: Device: Prevadh film
- Ringer solution (Active Comparator): Patients randomized in the Ringer solution group have been treated with Ringer lactate solution directly applied to the uterine surgical sites at the end of the myomectomy surgery.
  Interventions: Other: Ringer lactate solution

INTERVENTIONS:
Other: Ringer lactate solution — Ringer lactate solution was applied directly onto the uterine surgical sites at the end of the myomectomy surgery, to prevent post-surgical adhesion formation.
  Other Names: Myomectomy by Laparotomy
  Arms: Ringer solution
Device: Prevadh film — Prevadh film was applied directly onto the uterine surgical sites at the end of the myomectomy surgery to prevent post-surgical adhesion formation.
  Other Names: Myomectomy by Laparotomy
  Arms: Prevadh film

SUMMARY:
The purpose of this study was to evaluate clinically the efficacy of the PREVADH® Film in the prevention of adhesions in gynaecologic surgery, and to assess post-operative complications related to adhesions and pregnancy rate after myomectomy by open surgery.

DETAILED DESCRIPTION:
This study was addressed to patients having an immediate or differed pregnancy desire and presenting a symptomatic or asymptomatic fibroma being able to interfere with fertility.

* The primary end point was the assessment of adhesion rate to the uterine surgical sites during a laparoscopic second look performed 10 to 20 weeks post-surgery.
* The secondary end points were the assessment, throughout a 3 years follow-up period, of:

  * pregnancy rate,
  * adverse events related to adhesions,
  * adnexal adhesions according to American Fertility Society score,
  * abdomino-pelvic adhesions according to the modified American Fertility Society score.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic(s) or asymptomatic(s) uterin(s) fibroma(s) being able to interfere with the fertility by the patient who having an immediate or differed desire of pregnancy.
* Size: diameter ≥ 6 cm at echographia (for the highest diameter)
* Location interstitial and / or subserosa
* planned laparotomic surgery
* negative pregnancy test within 48 hours of surgery
* signed inform consent

Exclusion Criteria:

* History of abdomino-pelvic surgery (except appendicectomy - cesarotomy)
* Pre-operative embolization
* Endometriosis stage >1 (American Fertility Society classification ≥ 5)
* Pregnant patient
* Diabetes
* Chronic corticotherapy / immuno-supressor or immuno-modulator drugs
* Previous analog LH-RH drug therapy for the uterine myoma

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2006-05; Primary Completion 2008-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BECKER Patrice, Study Director — Sofradim Production; CANIS Michel, Pr, Principal Investigator — University Hospital Estaing - 63003 CLERMONT-FERRAND Cedex
Locations (11):
- France (11):
  - University Hospital, Angers
  - Clinique du Tondu, Bordeaux
  - Béclère Hospital (Public Assistance of Paris Hospital), Clamart
  - UNIVERSITY HOSPITAL Estaing, Clermont-Ferrand
  - University Carémeau Hospital, Nîmes
  - TENON Hospital (Public Assistance of Paris Hospital), Paris
  - TROUSSEAU Hospital (Public Assistance of Paris Hospital), Paris
  - Bichat Hospital - Claude Bernard (Public Assistance of Paris Hospital), Paris
  - South University Hospital, Rennes
  - Centre Hospitalier des quatre villes, Sèvres
  - Versailles Hospital, Versailles

REFERENCES:
- [Derived] Canis MJ, Triopon G, Darai E, Madelenat P, LeVeque J, Panel P, Fernandez H, Audebert A, Descamps P, Castaing N, Roman H, Fauconnier A, Benifla JL. Adhesion prevention after myomectomy by laparotomy: a prospective multicenter comparative randomized single-blind study with second-look laparoscopy to assess the effectiveness of PREVADH. Eur J Obstet Gynecol Reprod Biol. 2014 Jul;178:42-7. doi: 10.1016/j.ejogrb.2014.03.020. Epub 2014 Apr 8. PMID 24841647

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient included: 16 May 2006 Last patient included: 13 June 2008 11 participating centres, Hopsital
Groups:
- Prevadh™ (P) Group: Patients randomized in the Prevadh group have been treated with Prevadh film directly applied to the uterine surgical sites at the end of the myomectomy surgery.
- Ringer Lactate™ (R) Group: Patients randomized in the Ringer solution group have been treated with Ringer lactate solution directly applied to the uterine surgical sites at the end of the myomectomy surgery.
Period: Overall Study
Arm/Group | Prevadh™ (P) Group | Ringer Lactate™ (R) Group
Started | 33 | 28
Completed | 31 | 28
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prevadh™ (P) Group: Prevadh film was applied directly onto the uterine surgical sites at the end of the myomectomy surgery to prevent post-surgical adhesion formati.
- Total: Total of all reporting groups
Arm/Group | Prevadh™ (P) Group | Ringer Lactate™ (R) Group | Total
Number analyzed (Participants) | 33 | 28 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 28 | 61
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 33 | 28 | 61
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adhesions to Uterine Scars
Description: The primary endpoint was the assessment of adhesions to uterine scars and comprised the incidence (expressed per patient and per uterine scar), extent, and severity of adhesions observed during the second-look laparoscopy performed 10 to 20 weeks after the myomectomy.
  This assessment was made by the surgeon (investigator) on the one hand and by two independent surgeons who reviewed the video recordings on the other hand.
Time Frame: 10 to 20 weeks post surgery
Population: Two patients in group Prevadh group were withdrawn from the study, at 1 and 6 days post-myomectomy. One patient was re-operated for compress removal in Prevadh group and was excluded. Two patients in group Lactate Ringer group were withdrawn from the study, at 1 and 6 days post-myomectomy.
Measure: Number; unit: participants
Groups:
- Prevadh™ (P) Group: Prevadh film was applied directly onto the uterine surgical sites at the end of the myomectomy surgery to prevent post-surgical adhesion formation.
Arm/Group | Prevadh™ (P) Group | Ringer Lactate™ (R) Group
Number analyzed (Participants) | 28 | 26
participants | 12 | 24

2. Secondary Outcome: Fertility
Description: Fertility was assessed by pregnancy and deliveries rates at 3 years.
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Prevadh™ (P) Group | Ringer Lactate™ (R) Group
Number analyzed (Participants) | 28 | 26
participants
  Pregnancy rates at 3 years | 14 | 4
  Delivery rates at 3 years | 11 | 3

3. Secondary Outcome: Adnexal Adhesions
Description: Adnexal Adhesions were assessed by AFS score. AFS (= American Fertility Society) score was developed in 1980's by the American Fertility Society in an effort to address needs for a classification scheme for adnexal adhesions suspected to be associated with infertility. 4 anatomic sites evaluated: R-tube; R-ovary; L-tube; L-ovary. Final AFS score for a patient is the score of the side with lower summed score. The higher score, representing the side with the higher adhesion burden, is dropped; Score AFS is from 0 (best possible outcome) to 32 (worse possible outcome).
Time Frame: 10 to 20 weeks post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevadh™ (P) Group | Ringer Lactate™ (R) Group
Number analyzed (Participants) | 28 | 26
units on a scale | 4.0 (9.1) | 6.3 (12.2)

4. Secondary Outcome: mAFS Abdominopelvic Adhesion Score
Description: mAFS abdominopelvic adhesion score in 23 sites (at the anterior caudal peritoneum; parietocolic gutter right; right and left colon; right and left anterior cranial peritoneum; rectosigmoid; omentum; small intestine; anterior and posterior uterus; posterior cul-de-sac; right and left ovaries [internal and lateral sides], pelvic side walls, ovarian fossae, tubes, and bulbs). It ranges from 0 (best possible outcome) to 16 (worse possible outcome).
Time Frame: 10 to 20 weeks post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevadh™ (P) Group | Ringer Lactate™ (R) Group
Number analyzed (Participants) | 28 | 26
units on a scale | 1.6 (2.7) | 2.4 (3.5)

ADVERSE EVENTS:
Groups:
- Prevadh™ (P) Group With Adverse Event: Patients randomized in the Prevadh group have been treated with Prevadh Film directly applied to the uterine surgical sites at the end of the myomectomy surgery.
- Ringer Lactate™ (R) Group With Adverse Event: Patients randomized in the Ringer solution group have been treated with Ringer lactate solution directly applied to the uterine surgical sites at the end of the myomectomy surgery.
  .
Arm/Group | Prevadh™ (P) Group With Adverse Event | Ringer Lactate™ (R) Group With Adverse Event
Serious Adverse Events (participants affected / at risk) | 7/33 | 4/28
Other Adverse Events (participants affected / at risk) | 9/33 | 7/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevadh™ (P) Group With Adverse Event (N=33) | Ringer Lactate™ (R) Group With Adverse Event (N=28)
Achilles tendon rupture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Miscarriage on first quarter/SAE due to deliveries (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
ovarian hyperstimulation and in vitro fertilization (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
intra-abdominal bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anemia due to pre- and post-operative bleeding (metrorragia) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Parietal hematoma requiring Hospitalization (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abdominal pain and digestive disorders/SAE due to deliveries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Compress removal/Small intestine's adhesions, requiring hospitalization (Surgical and medical procedures) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Submucosal myoma requiring re-intervention (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Intra-uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevadh™ (P) Group With Adverse Event (N=33) | Ringer Lactate™ (R) Group With Adverse Event (N=28)
Calf Pain (negative Doppler for phlebitis) (Vascular disorders) | 1 (1) | 0 (0)
Varicella AND Parietal hematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Continuous pelvic pain AND Mild separation of the parietal scar (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Thoracic Pain (negative angioscanner) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Superficial injury of sigmoid during coelioscopy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fever during 48-hours post-surgery (Infections and infestations) | 0 (0) | 1 (1)
Keloid laparoscopic scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hemorrhagic uterus during myomectomy (Reproductive system and breast disorders) | 0 (0) | 1 (1)
38.8°C Fever (Infections and infestations) | 1 (1) | 0 (0)
Submucosal myoma (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Metrorragia due to uterine cavity opening. (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Parietal hematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematoma on umbilical scar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fever (38.5°C) (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
the surgeons were not blinded to the patients' allocation group at second-look laparoscopy.Recruitment was stopped early. 2 data analyses have been performed over the study period for primary endpoint, without any error type I adjustment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less